CLINICAL TRIAL: NCT04589702
Title: Temporal Activation of Core Muscles and Vasti in Isolated Patellofemoral Osteoarthritis During Stair-stepping
Brief Title: Temporal Activation of Core Muscles and Vasti in Isolated Patellofemoral Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, afaf mohamed omar tahoon, assistant lecturer, Cairo University
Other Study IDs: (P.T.Rec/012/001659)
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chondromalacia Patellae
MeSH Terms: conditions — Chondromalacia Patellae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- females with isolated patellofemoral arthritis: those with anterior knee pain
- healthy females: those without anterior knee pain

SUMMARY:
Objective: To compare the temporal muscle activation between females with PF OA and normal controls during stair ascent. Methods: An observational comparative study was conducted with thirty-one females with PF OA and 11 healthy ones. The onset times of multifidus, transversus abdominus (TrA), gluteus medius (GM), and vasti muscles were measured by quantitative Electromyography during stair ascent task. hypothesis: Investigators hypothesized that there won't be a significant difference between females with PF OA and their matched healthy group regarding the onset times of vastus medialis obliqus (VMO), vastus lateralis (VL), gluteus medius (GM), multifidus, and transversus abdominus (TrA), during stair ascent task.

DETAILED DESCRIPTION:
Investigators collected the EMG activity of VMO, VL, GM, multifidus, and TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada). Electromyographic data were sampled at 1000 Hz and bandpass filtered at 50-200 Hz.

For each muscle, three electrodes were used; two electrodes were placed ~ 30 mm apart in the direction of the muscle fibers and a ground electrode was placed over the closest bony prominence. Before placement of the electrodes, the subject's skin was cleaned with alcohol to reduce impedance and excess hair was removed to eliminate shifting of the electrodes if needed.

The stair-stepping task consisted of ascending 2 steps (each step was 40 cm in width, 20 cm in height, without handrails. The depth of the first and second steps was 30 cm and 40 cm, respectively) . Participants were asked to stand on the floor confronting the stairs and 20 cm away from the edge of the initial step. The stair ascent task was performed barefooted while arms hanged at the side of the body. Patients started ascending the steps immediately in response to a command, at their normal speed with their affected limb. Investigators didn't control the speed of stair ascent, because controlling the timing of stair-stepping can alter the electromyographic signal as shown earlier for gait in asymptomatic subjects. Healthy subjects started ascending stairs with their dominant limb .

Before data acquisition, participants performed one practice trial of stair ascent to get familiarized with the task. Then the participants performed three test trials with thirty seconds of rest after each trial to prevent fatigue. The raw data were stored on a personal computer for analysis with a custom program in Matlab (Math Works, Natick, Massachusetts, USA). Investigators used a mean of data in three trials for analysis.

Statistical Analysis:

Data management and analysis were conducted using the statistical package for social studies (SPSS) version 22 for windows (IBM SPSS, Chicago, IL, USA). Normal distribution of the data was tested using the Shapiro-Wilk test. The homogeneity of variances between groups was examined using Levene's test. Descriptive data are expressed as mean ± standard deviation. An independent t-test was conducted for comparison of subject characteristics; age, body mass index (BMI), weight and height, between both groups. A univariate test of one way MANOVA was performed to compare EMG onset of each muscle between both groups. Post-hoc analysis using the Bonferroni method was carried out for subsequent multiple comparison. The level of significance for all statistical tests was set at p < 0.05.

ELIGIBILITY:
* Inclusion Criteria for PF OA group; patients included if they had

  1. Anterior- or retro-patellar knee pain aggravated by at least two activities that load the PFJ (eg; stair ambulation, squatting and/or rising from sitting) .
  2. Pain during these activities presented on most days during the past month and their pain severity was ≥ 4 on an 11 point numerical pain scale during aggravating activities .,
  3. A grade less than (2) from postero-anterior views on the Kellgren - Lawrence (KL) grading scale.
* Inclusion Criteria for Healthy control subjects :

  1. no history of knee pathology or pain with any of the provocative activities which were mentioned above.
* Exclusion Criteria for Patients in the PF OA group:

  1. concomitant pain from tibiofemoral joint or other knee structures .
* Exclusion Criteria for Subjects from both groups:

  1. current or previous pain in the hip, lumbar spine or foot that had lasted longer than 3 months and/or required intervention.
  2. a history of lower extremity, pelvis or spine fractures; spine, hip, knee or foot surgeries; hip or patellar subluxation/ dislocation.
  3. injury to any of knee ligaments or meniscus.
  4. systemic diseases (e.g. rheumatoid arthritis), neurological conditions or fibromyalgia . 5.The professional athletes; people who exercise more than two hours a day or every other day, were also excluded .

     -

Ages: 35 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Patients were recruited from the Outpatient Clinic of Kasr Al-Ainy Hospital and the Faculty of Physical Therapy, Cairo University as well. However, control subjects were recruited via advertising in the local community.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The EMG onset of multifidus, transversus abdominus (TrA), gluteus medius (GM), and vasti muscles | from admission to discharge, up to two weeks
  investigators collected the EMG activity of VMO, VL, GM, multifidus, and TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).

CONTACTS AND LOCATIONS:
Overall Officials: Aladdin A. balbaa, professor, Study Director — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No